CLINICAL TRIAL: NCT03519594
Title: The Size of Pelvic Hematoma Can be a Predictive Factor for Angioembolization in Hemodynamically Unstable Pelvic Trauma
Brief Title: The Size of Pelvic Hematoma Can be a Predictive Factor for Angioembolization
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Suk-Kyung, Associate professor, Asan Medical Center
Other Study IDs: AsanMC-Hematoma
Record Dates: First submitted 2018-04-20; First posted 2018-05-09 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Multiple Pelvic Fractures
Keywords: angioembolization; computed tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Embolization group: The group that underwent embolization after pelvic injury.
- Non-embolization group: The observed group of pelvic injuries without embolization

SUMMARY:
Unstable pelvic fracture with bleeding can be fatal, with a mortality rate of up to 40%. Therefore, early detection and treatment are important in unstable pelvic trauma. We investigated the early predictive factors for possible embolization in patients with hemodynamically unstable pelvic trauma. The purpose of this study was to predict the necessity of embolization and the timing of angiography using CT scans.

DETAILED DESCRIPTION:
Background: Unstable pelvic fracture with bleeding can be fatal, with a mortality rate of up to 40%. Therefore, early detection and treatment are important in unstable pelvic trauma. We investigated the early predictive factors for possible embolization in patients with hemodynamically unstable pelvic trauma.

Methods: From January 2011 to December 2013, 46 patients with shock arrived at a single hospital within 24 h after injury. Of them, 44 patients underwent computed tomography (CT) after initial resuscitation, except for 2 who were dead on arrival. Nine patients with other organ injuries were excluded. Seventeen patients underwent embolization. A single radiologist measured the width (longest length in axial view) and length (longest length in coronal view) of pelvic hematoma on CT scans. Demographic, clinical, and radiological data were reviewed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* patients with shock (systolic blood pressure <90 mmHg) arrived at a single hospital within 24 h after injury after pelvic fracture

Exclusion Criteria:

* declared dead on arrival
* patients with other organ injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with major trauma and pelvic bone fracture
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Predictive factors for embolization in unstable pelvic fracture | 2 years
  The factors affecting embolization are analyzed by logistic regression analysis

SECONDARY OUTCOMES:
The odds ratio of mortality rate between two groups | 2 years
  Obtain the difference in mortality rate between two groups
Cut-off values of pelvic hematoma width | 2 years
  Measure the length of pelvic hematoma using the ROC curve

CONTACTS AND LOCATIONS:
Overall Officials: Suk-kyung Hong, Ph.D., Principal Investigator — Asan Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coccolini F, Stahel PF, Montori G, Biffl W, Horer TM, Catena F, Kluger Y, Moore EE, Peitzman AB, Ivatury R, Coimbra R, Fraga GP, Pereira B, Rizoli S, Kirkpatrick A, Leppaniemi A, Manfredi R, Magnone S, Chiara O, Solaini L, Ceresoli M, Allievi N, Arvieux C, Velmahos G, Balogh Z, Naidoo N, Weber D, Abu-Zidan F, Sartelli M, Ansaloni L. Pelvic trauma: WSES classification and guidelines. World J Emerg Surg. 2017 Jan 18;12:5. doi: 10.1186/s13017-017-0117-6. eCollection 2017. PMID 28115984
- [Result] Hymel A, Asturias S, Zhao F, Bliss R, Moran T, Marshall RH, Benjamin E, Phelan HA, Krause PC, Marecek GS, Leonardi C, Stuke L, Hunt JP, Mooney JL. Selective versus nonselective embolization versus no embolization in pelvic trauma: A multicenter retrospective cohort study. J Trauma Acute Care Surg. 2017 Sep;83(3):361-367. doi: 10.1097/TA.0000000000001554. PMID 28463936
- [Result] Salim A, Teixeira PG, DuBose J, Ottochian M, Inaba K, Margulies DR, Demetriades D. Predictors of positive angiography in pelvic fractures: a prospective study. J Am Coll Surg. 2008 Nov;207(5):656-62. doi: 10.1016/j.jamcollsurg.2008.05.025. Epub 2008 Jul 14. PMID 18954776
- [Result] Blackmore CC, Cummings P, Jurkovich GJ, Linnau KF, Hoffer EK, Rivara FP. Predicting major hemorrhage in patients with pelvic fracture. J Trauma. 2006 Aug;61(2):346-52. doi: 10.1097/01.ta.0000226151.88369.c9. PMID 16917449